CLINICAL TRIAL: NCT05581277
Title: Efficacy of the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders (UP) in People With Post Covid-19 Condition and Emotional Symptomatology.
Brief Title: Efficacy of the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders (UP) in People With Post Covid-19 Condition.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PUCPCovid
Record Dates: First submitted 2022-10-13; First posted 2022-10-14 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2022-10

CONDITIONS: Emotional Disorder; Post COVID-19 Condition; Anxiety Disorders; Depressive Disorder
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder

STUDY DESIGN:
Intervention Model Description: In the present investigation, all consecutive patients presenting post covid-19 condition and symptoms of anxiety or depression are requested to participate. Once inclusion criteria are accomplished, each patient will be randomly assigned to one of the multiple baseline groups: 6, 8 or 10 days of assessment before the intervention. The study includes seven assessment points (baseline, pre-treatment, post-treatment and four follow-ups, at one, three, six and twelve months after completion of treatment).
Who Masked: Participant
Masking Description: Participants will know the baseline condition they have been assigned to: 6, 8 or 10 evaluation days before the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Comparator: 6 days before intervention (Active Comparator): Participants have to complete a pre-treatment assessment (baseline) for 6 days.
  Interventions: Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders
- Active Comparator: 8 days before intervention (Active Comparator): Participants have to complete a pre-treatment assessment (baseline) for 8 days.
  Interventions: Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders
- Active Comparator: 10 days before intervention (Active Comparator): Participants have to complete a pre-treatment assessment (baseline) for 10 days.
  Interventions: Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders

INTERVENTIONS:
Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders — This intervention focuses on a wide range of emotional psychopathology, allowing care for comorbid disorders and subclinical or unspecified symptoms, which reduces treatment times and costs, and improves response to treatment. The intervention will be carried out in an online-individual format.

SUMMARY:
The present multiple baseline single case trial will study the efficacy and acceptability of the "Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders" in the treatment of emotional symptomatology and/or emotional disorders in a sample of patients with Post Covid-19 condition.

DETAILED DESCRIPTION:
COVID-19 disease has caused one of the largest pandemics in world history. Two and a half years after the WHO declared a pandemic status for COVID-19, it is known that about 10-20% of Covid-19 patients fail to recover their initial health status and report persistent symptoms over time. This group of people suffer from what has been defined by the WHO as post-COVID-19 condition. Among this group of patients, the most common symptoms observed are fatigue, shortness of breath and cognitive dysfunction, as well as psychological sequelae. Among the latter, the group of Emotional Disorders ( EDs), a nomenclature that groups anxiety disorders, depressive and related disorders, are those most commonly reported by people with post-COVID-19 condition, with alarmingly high rates of persistent psychological distress (36%), anxiety disorders (22%), depression (21%), post-traumatic stress disorder (20%) and sleep disorders (35%). Therefore, it is necessary to apply intervention programs for the treatment of psychological sequelae derived from post-COVID-19 condition, as well as emotional demands and needs in this population highly affected by the COVID-19 pandemic.

The overall objective of this trial is to study the efficacy and acceptability of the "Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders" (UP) in the treatment of emotional symptomatology and/or ED in a sample of patients with post-COVID-19 condition. The investigators hypothesize that a structured psychological intervention focused on treating emotional dysregulation (the UP), a factor shared by the group of EDs, will generate an improvement in the emotional state of this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Belong to the autonomous community of Aragón
* Be at least 18 years of age
* Have a good understanding of Spanish
* SARS CoV 2 infection documented by PCR, Ag test or serology
* Persistence of symptoms beyond 12 weeks after acute SARS CoV 2 infection
* Emotional symptoms (score equal to or greater than 8 points in anxious symptomatology(OASIS) and/or equal to or greater than 7 points in depressive symptomatology (ODSIS)) and/or diagnosis of Emotional disorder (ED)
* Internet access available
* Signed informed consent.

Exclusion Criteria:

* Participating in the trial "Specialized nutritional intervention and rehabilitative treatment for improvement of quality of life in a cohort of patients with post covid-19 condition"
* That the symptom(s) already existed prior to acute SARS CoV 2 infection
* Receiving psychological and/or pharmacological treatment for a mental disorder at present
* Having a diagnosis of severe mental disorder
* Active suicidal ideation at the time of evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Sociodemographic data | Pre-treatment
  sex, age, place of residence (zip code), marital status, employment status, lifestyle habits (smoking, alcohol, physical activity, diet), SARS CoV 2 vaccination (Yes/No prior to infection, number and date of doses, brand of vaccine)
Table of symptoms referred by the patient | Up to 12 months
  To facilitate the collection of symptoms referred by the patient regarding CPCOVID, we have developed a table in which different symptoms present in this condition are collected, grouped into the following categories: General Symptoms, Respiratory Symptoms, Gastrointestinal Symptoms, Musculoskeletal Symptoms, Cutaneous Symptoms, Otolaryngological Symptoms, Neurological Symptoms, Cardiovascular Symptoms, Psychological Symptoms and Others
Overall Anxiety Severity and Impairment Scale (OASIS) | Up to 12 months
  Consist of five items that evaluate the frequency and the intensity of anxious symptoms and their interference with the person's work or school life and social life. The total score range from 0 to 20 and responses use a 5-point Likert scale ranging from 0 to 4. Higher scores are indicative of greater severity and functional impairment as a result of anxious symptoms.
Overall Depression Severity and Impairment Scale (ODSIS) | Up to 12 months
  Consist of five items that evaluate the frequency and the intensity of depressive symptoms and their interference with the person's work or school life and social life. The total score range from 0 to 20 and responses use a 5-point Likert scale ranging from 0 to 4. Higher scores are indicative of greater severity and functional impairment as a result of depressive symptoms.
Anxiety and related disorders interview (ADIS-5) | Pre-treatment
  Structured interview following DSM-5 criteria for anxiety, mood and related disorders
Adjustment disorders | Pre-treatment
  Adjustment disorders will be evaluated according to DSM-5 criteria.

SECONDARY OUTCOMES:
The Multidimensional Emotional Disorder Inventory (MEDI) | Up to 12 months
  A self-report measure that includes only 49 items and enables to quickly assess the main transdiagnostic dimensions of Emotional disorders
Health-related quality of life (EuroQol-5D) | Up to 12 months
  Evaluation through 5 items of quality of life.
Difficulties in Emotion Regulation Scale (DERS) | Up to 12 months
  Consists of 36-item of six facets of emotion regulation. Items are rated on a scale of 1 ("almost never [0-10%]") to 5 ("almost always [91-100%]"). Higher scores indicate more difficulty in emotion regulation
Distress Tolerance Scale (DTS) | Up to 12 months
  Assessment through 15 items of distress tolerance
Adaptation of Client Satisfaction Questionnaire [CSQ-8] | Up to 12 months
  An adaptation of 7 items that measures quality of the intervention and its components, discomfort experienced during treatment and the experience of participating in an online individual format.
Evaluation questionnaire of the Unified Protocol (UP) modules | Up to 12 months
  Consists of 7 items that evaluate the usefulness of the program to improve emotional regulation and the usefulness of each of the skills that are worked on in the different UP modules
Baseline assessment questionnaire | Up to 12 months
  For the daily baseline assessment, we will use the ODSIS and OASIS questionnaires by modifying the temporality to which the questions refer; changing from "during the last week" in the original questionnaires to "during yesterday" in the version used for the baseline assessment

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Lozano Blesa Clinical University Hospital, Zaragoza, Aragon
  - Jorge Osma, Teruel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinez-Borba V, Martinez-Garcia L, Peris-Baquero O, Osma J, Del Corral-Beamonte E. Unified Protocol for the transdiagnostic treatment of emotional disorders in people with post COVID-19 condition: study protocol for a multiple baseline n-of-1 trial. Front Psychol. 2023 Oct 18;14:1160692. doi: 10.3389/fpsyg.2023.1160692. eCollection 2023. PMID 37920733